CLINICAL TRIAL: NCT01635985
Title: A Phase I, Single Centre, Open, Partly Randomised, Crossover Study in Healthy Subjects to Evaluate AZD5423 Absolute Pulmonary Bioavailability When Administered Inhaled Via a New Dry Powder Inhaler, Turbuhaler, Spira Nebulizer and I-neb AAD System
Brief Title: A Study in Healthy Subjects to Investigate Pharmacokinetics of AZD5423 When Administered in Different Ways
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D2340C00012; Eudract 2012-002307-17
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Bioavailability and AUC
Keywords: Phase I, Healthy male volunteers, pharmacokinetics
MeSH Terms: interventions — 2,2,2-trifluoro-N-(1-((1-(4-fluorophenyl)-1H-indazol-5-yl)oxy)-1-(3-methoxyphenyl)-2-propanyl)acetamide

ARMS (6):
- 1 (Experimental): AZD5423 iv
  Interventions: Drug: AZD5423
- 2 (Experimental): AZD5423 inhalation, Spira
  Interventions: Drug: AZD5423
- 3 (Experimental): AZD5423 inhalation I-neb
  Interventions: Drug: AZD5423
- 4 (Experimental): AZD5423 oral
  Interventions: Drug: AZD5423
- 5 (Experimental): AZD5423 inhalation Turbuhaler
  Interventions: Drug: AZD5423
- 6 (Experimental): AZD5423, New Dry Powder Inhaler
  Interventions: Drug: AZD5423

INTERVENTIONS:
Drug: AZD5423 — solution for injection, administered as intravenous infusion Corr to total dose of 250 µg AZD5423
  Arms: 1
Drug: AZD5423 — nebuliser suspension, inhaled via Spira, corr to approximately 300 µg lung deposited dose AZD5423
  Arms: 2
Drug: AZD5423 — nebuliser suspension, inhaled via I-neb, corr to approximately 300 µg lung deposited dose AZD5423
  Arms: 3
Drug: AZD5423 — nebuliser suspension to be administered orally, corr to a total dose of 1200 µg AZD5423
  Arms: 4
Drug: AZD5423 — dry powder inhaled via Turbuhaler, corr to approximately 200 µg lung deposited dose AZD5423
  Arms: 5
Drug: AZD5423 — dry powder inhaled via New Dry Powder Inhaler, corr to approximately 200 µg lung deposited dose AZD5423
  Arms: 6

SUMMARY:
The purpose of this study is to look at drug levels of AZD5423 in blood when the drug is administered in different ways - orally, intravenously or inhaled (with four different devices), to healthy subjects

DETAILED DESCRIPTION:
A Phase I, Single Centre, Open, Partly Randomised, Crossover Study in Healthy Subjects to Evaluate AZD5423 Absolute Pulmonary Bioavailability when Administered Inhaled via a New Dry Powder Inhaler, Turbuhaler, Spira nebulizer and I-neb AAD system

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or women of non-childbearing potential aged 18-45 years inclusive with suitable veins for cannulation or repeated vein puncture
* Have a body mass index (BMI) between 19 and 30 kg/m2 (inclusive and rounding allowed) and weight between 50 and 100 kg (inclusive)
* Be able to inhale from the inhaler devices used in the study according to given instructions as well as be able to perform spirometry

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Current smokers
* Any clinically relevant abnormal findings

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of AZD5423 delivered by the new dry powder inhaler in terms of: Fpulmonary | Blood samples taken pre-dose and at10, 20 and 40 minutes and 1, 1.5, 2, 4, 6, 8, 12,16, 24, 36, 48 and 96 hours post dose.

SECONDARY OUTCOMES:
Pharmacokinetics of AZD5423 following i.v administration in terms of : AUC, AUC(0-t), Fpo, Finhalation total, Fpulmonary, Foral, Frel, Frel Cmax, Cmax, Cmax(tmax), t½λz, MAT, MRT, Vz and Vss | Blood samples taken pre-dose and at 5, 10, 25, 30, 35 and 45 minutes and 1, 1.5, 2, 4, 6, 8, 12,16, 24, 36, 48, 72 and 96 hours post dose.
Pharmacokinetics of AZD5423 following oral administration in terms of : AUC, AUC(0-t), Fpo, Finhalation total, Fpulmonary, Foral, Frel, Frel Cmax, Cmax, Cmax(tmax), t½λz, MAT, MRT, Vz and Vss | Blood samples taken pre-dose and at10, 20 and 40 minutes and 1, 1.5, 2, 4, 6, 8, 12,16, 24, 36 and 48 hours post dose.
Pharmacokinetics of AZD5423 following oral inhalation by Spira, I-neb, Turbuhaler and New Dry Powder Inhaler in terms of : AUC, AUC(0-t), Fpo, Finhalation total, Fpulmonary, Foral, Frel, Frel Cmax, Cmax, Cmax(tmax), t½λz, MAT, MRT, Vz and Vss | Blood samples taken pre-dose and at10, 20 and 40 minutes and 1, 1.5, 2, 4, 6, 8, 12,16, 24, 36, 48 and 96 hours post dose.
Safety profile in terms of adverse events, ECG, heart rate, blood pressure, pulse rate, body temperature, physical examination, spirometry, haematology, clinical chemistry and urinalysis. | Screening to 28 days post dose.
  No formal statistical tests will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, MD, Study Director — AstraZeneca R&D, Molndal Sweden
Locations (1):
- London, UK, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1259&filename=D2340C00012.pdf